CLINICAL TRIAL: NCT03599089
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Safety, Pharmacokinetics and Efficacy Study of CA-008 in Subjects Undergoing Bunionectomy
Brief Title: Study of CA-008 (Vocacapsaicin) in Bunionectomy Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Concentric Analgesics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA-PS-201
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Post-surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ketorolac; Acetaminophen; Oxycodone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CA-008 (vocacapsaicin) 0.7 mg (0.05 mg/mL concentration) (Active Comparator): Each patient will receive a single dose of 0.7 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone; Drug: Bupivacaine Hydrochloride
- CA-008 (vocacapsaicin) 2.1 mg (0.15 mg/mL concentration) (Active Comparator): Each patient will receive a single dose of 2.1 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone; Drug: Bupivacaine Hydrochloride
- CA-008 (vocacapsaicin) 4.2 mg (0.3 mg/mL concentration) (Active Comparator): Each patient will receive a single dose of 4.2 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  Interventions: Drug: CA-008; Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone; Drug: Bupivacaine Hydrochloride
- Placebo (Placebo Comparator): Each patient will receive a single dose of CA-008 vehicle (identical to active treatment but without CA-008) injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  Interventions: Drug: Placebo; Drug: Ketorolac; Drug: Acetaminophen; Drug: Oxycodone; Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: CA-008 — single-dose wound infiltration prior to surgical incision closure
  Other Names: Vocacapsaicin
  Arms: CA-008 (vocacapsaicin) 0.7 mg (0.05 mg/mL concentration); CA-008 (vocacapsaicin) 2.1 mg (0.15 mg/mL concentration); CA-008 (vocacapsaicin) 4.2 mg (0.3 mg/mL concentration)
Drug: Placebo — single-dose wound infiltration prior to surgical incision closure
  Arms: Placebo
Drug: Ketorolac — 30mg IV administered intraoperatively
Drug: Acetaminophen — 1000mg IV administered intraoperatively
Drug: Oxycodone — 5mg PO prn post-surgery
Drug: Bupivacaine Hydrochloride — 0.5% infiltration pre-surgery

SUMMARY:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, parallel design study evaluating a single dose of one of three CA-008 dose levels vs. placebo injected during an elective bunionectomy Bunionectomy to assess post-surgical pain management and the need for rescue medication (oxycodone).

DETAILED DESCRIPTION:
Primary Objective:

To evaluate the efficacy of a single intraoperative administration of CA- 008 vs placebo in subjects undergoing an elective Bunionectomy .

Secondary Objectives

* To evaluate the safety and tolerability of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective Bunionectomy.
* To evaluate the PK profile of a single intraoperative administration of CA-008 vs. placebo in subjects undergoing an elective Bunionectomy .
* To explore the efficacy of various doses of CA-008 administered intraoperatively in subjects undergoing an elective Bunionectomy .

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged 18 - 75 years old
2. American Society of Anesthesiology (ASA) physical Class 1, 2 or 3
3. Planning elective Bunionectomy repair
4. For both males and females: using an acceptable method of birth control
5. If a female: not pregnant or breastfeeding
6. Have a body mass index ≤ 40 kg/m2.
7. Be willing and able to sign the informed consent form (ICF)
8. Be able to complete study procedures and pain scales and to communicate meaningfully in English
9. Be willing to undergo 17 blood draws for pharmacokinetic (PK )assessments over 24 hours

Exclusion Criteria:

1. Have another painful condition, other than bunion-related pain, that may require pain treatment during the study period
2. Have active skin disease or another abnormality at the anticipated site of surgery that could interfere with the planned surgery.
3. Have a known allergy to chili peppers, capsaicin or the components of CA-008, bupivacaine HCl, ketorolac, acetaminophen or oxycodone.
4. Have a history of significant medical, neuropsychiatric or other condition, including a clinically significant abnormal clinical laboratory test values
5. Be on any medication not allowed per the protocol
6. Within the past year have a history of illicit drug use or prescription medicine or alcohol abuse
7. Have positive results on the alcohol test (breath or saliva) or urine drug screen
8. Have previously participated in a clinical study with CA-008.
9. Have participated in another clinical trial or used an investigational product within 30 days or five half-lives (whichever is longer)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Wu, Study Director — Concentric Analgesics
Locations (3):
- United States (3):
  - Lotus Clinical Research, LLC, Pasadena, California
  - Chesapeake Research Group, Pasadena, Maryland
  - HD Research Corp, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- CA-008 0.7 mg (0.05 mg/mL Concentration): Each patient will receive a single dose of 0.7 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  CA-008: single-dose wound infiltration prior to surgical incision closure
  Ketorolac: 30mg IV administered intraoperatively
  Acetaminophen: 1000mg IV administered intraoperatively
  Oxycodone: 5mg PO prn post-surgery
  Bupivacaine Hydrochloride: 0.5% infiltration pre-surgery
- CA-008 2.1 mg (0.15 mg/mL Concentration): Each patient will receive a single dose of 2.1 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  CA-008: single-dose wound infiltration prior to surgical incision closure
  Ketorolac: 30mg IV administered intraoperatively
  Acetaminophen: 1000mg IV administered intraoperatively
  Oxycodone: 5mg PO prn post-surgery
  Bupivacaine Hydrochloride: 0.5% infiltration pre-surgery
- CA-008 4.2 mg (0.3 mg/mL Concentration): Each patient will receive a single dose of 4.2 mg CA-008 injected during an elective Bunionectomy with a multimodal analgesia regimen including a Nonsteroidal anti-inflammatory drug (NSAID) and regional Mayo block with bupivacaine.
  CA-008: single-dose wound infiltration prior to surgical incision closure
  Ketorolac: 30mg IV administered intraoperatively
  Acetaminophen: 1000mg IV administered intraoperatively
  Oxycodone: 5mg PO prn post-surgery
  Bupivacaine Hydrochloride: 0.5% infiltration pre-surgery
Period: Overall Study
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo
Started | 36 | 36 | 38 | 37
Completed | 33 | 35 | 37 | 35
Not Completed | 3 | 1 | 1 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo | Total
Number analyzed (Participants) | 36 | 36 | 38 | 37 | 147
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.29) | 44.6 (12.33) | 41.4 (12.16) | 50.7 (12.46) | 46.4 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 25 | 34 | 31 | 123
  Male | 3 | 11 | 4 | 6 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 11 | 8 | 12 | 39
  Not Hispanic or Latino | 28 | 25 | 30 | 25 | 108
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 0 | 2
  Asian | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1 | 2
  Black or African American | 12 | 12 | 14 | 14 | 52
  White | 20 | 20 | 19 | 22 | 81
  More than one race | 3 | 3 | 2 | 0 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 36 | 36 | 38 | 37 | 147

OUTCOME MEASURES:

1. Primary Outcome: Change in Postsurgical Pain Based on the Weighted Sum of Pain Intensity (SPI) Assessments Over 96 Hours of the NRS Scores = Area Under the Curve (AUC)
Description: Mean area under the curve (AUC) of the Numeric Rating Scale (NRS) weighted sum of pain intensity scores (at rest) from 0-10 where 0 is no pain and 10 is the worst pain imaginable for CA-008 compared to placebo. The time was collected 0 to 96 hours post-dose
Time Frame: [time frame: 96 hours]
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: scores on a scale*hour
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo
Number analyzed (Participants) | 36 | 36 | 38 | 37
scores on a scale*hour | 317.09 (204.291) | 321.72 (165.145) | 266.86 (220.674) | 400.56 (215.471)
Statistical Analysis 1: Comparison: CA-008 4.2 mg (0.3 mg/mL Concentration) vs Placebo; Test type: Superiority; p = 0.005, ANOVA

2. Secondary Outcome: Percentage of Subjects Opioid Free
Description: Percentage of subjects who are opioid-free for CA-008 compared to placebo.
Time Frame: [time frame: 96 hours]
Population: Modified Intent to Treat
Measure: Number; unit: percentage of subjects
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo
Number analyzed (Participants) | 36 | 36 | 38 | 37
percentage of subjects | 19.4 | 16.7 | 26.3 | 5.4
Statistical Analysis 1: Comparison: CA-008 4.2 mg (0.3 mg/mL Concentration) vs Placebo; Test type: Superiority; p = 0.0245, Regression, Logistic

3. Secondary Outcome: Total Opioid Consumption (in Daily Morphine Equivalents)
Description: Mean total postoperative opioid consumption (in daily oral morphine equivalents) for CA-008 compared to placebo
Time Frame: [time frame: 96 hours]
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: mg morphine equivalents/day
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo
Number analyzed (Participants) | 36 | 36 | 38 | 37
mg morphine equivalents/day | 42.50 (38.074) | 37.71 (39.340) | 28.22 (28.355) | 56.11 (45.447)
Statistical Analysis 1: Comparison: CA-008 4.2 mg (0.3 mg/mL Concentration) vs Placebo; Test type: Superiority; p = 0.0019, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time that each participant provided written informed consent (up to 45-day screening period) through Day 36+2 days. The total duration could be a maximum of 83 days.
Arm/Group | CA-008 0.7 mg (0.05 mg/mL Concentration) | CA-008 2.1 mg (0.15 mg/mL Concentration) | CA-008 4.2 mg (0.3 mg/mL Concentration) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/36 | 0/38 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 0/38 | 1/37
Other Adverse Events (participants affected / at risk) | 27/36 | 28/36 | 26/38 | 25/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 0.7 mg (0.05 mg/mL Concentration) (N=36) | CA-008 2.1 mg (0.15 mg/mL Concentration) (N=36) | CA-008 4.2 mg (0.3 mg/mL Concentration) (N=38) | Placebo (N=37)
Cellulitis on left big toe (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CA-008 0.7 mg (0.05 mg/mL Concentration) (N=36) | CA-008 2.1 mg (0.15 mg/mL Concentration) (N=36) | CA-008 4.2 mg (0.3 mg/mL Concentration) (N=38) | Placebo (N=37)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 1 (1) | 4 (4)
Nausea (Gastrointestinal disorders) | 6 (6) | 7 (7) | 7 (7) | 9 (9)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4) | 3 (3) | 4 (4)
Feeling hot (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Infusion site oedema (General disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 3 (3) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 7 (7) | 8 (8) | 7 (7) | 6 (6)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin maceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood pressure increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye haematoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Administration site warmth (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Application site rash (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion site pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incision site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diastolic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT03599089/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-09): https://cdn.clinicaltrials.gov/large-docs/89/NCT03599089/SAP_001.pdf